CLINICAL TRIAL: NCT01368809
Title: Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Effect of Fentanyl on the Incidence of Coughing and Recovery After Propofol-Desflurane Anesthesia With an LMA for Airway Management
Brief Title: Effect of Fentanyl on Coughing and Recovery After Anesthesia With an LMA Laryngeal Mask Airway)for Airway Management
Acronym: LMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ronald Wender, Chairman, Department of Anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00024484
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Ambulatory Surgery; Coughing
Keywords: Ambulatory surgery; Pain management; Perioperative outcomes; Fentanyl; Coughing during insertion of an LMA; Ambulatory surgery procedures
MeSH Terms: conditions — Cough; Agnosia | interventions — Sodium Chloride; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl (Active Comparator): Fentanyl (50 µg/ml) 2 ml at induction, 1-2 ml boluses as needed
  Interventions: Drug: Fentanyl
- Saline Solution (Placebo Comparator): Saline Solution 2 ml at induction, 1-2 ml boluses as needed
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — 2 ml at induction 1-2 ml boluses as needed
  Other Names: placebo
  Arms: Saline Solution
Drug: Fentanyl — Fentanyl (50 µg/ml) 2 ml at induction, 1-2 ml boluses as needed
  Arms: Fentanyl

SUMMARY:
The purpose of this research is to evaluate the effectiveness of fentanyl for reducing coughing during the perioperative period (i.e., insertion of an LMA [Laryngeal Mask Airway] device, maintenance period during surgery, and awakening [emergence] from general anesthesia) for ambulatory surgery procedures. Also to assess the effects of fentanyl on the postoperative outcomes, (e.g., pain, postoperative nausea and vomiting, return of bowel function [constipation], resumption of normal activities of daily living).

Fentanyl is one of the most common used anesthetic adjuncts for ambulatory surgery because of its anesthetic-sparing effects and alleged ability to reduce coughing during instrumentation of the patient's airway.

DETAILED DESCRIPTION:
This research study is designed to evaluate the effects of fentanyl when administered as an adjuvant to standard anesthetic and analgesic drugs on coughing (during insertion of an LMA device, during maintenance and emergence from general anesthesia) and on the postoperative adverse outcomes (i.e., side effects).

All patients will receive local anesthetics and commonly used non-opioid pain relieving medications during surgery.

ELIGIBILITY:
Inclusion Criteria

* Patients scheduled to undergo outpatient arthroscopic surgery procedures
* Willingness and ability to sign an informed consent document
* No allergies to anesthetic or analgesic medications
* 18 - 80 years of age
* American Society of Anesthesiologists (ASA) Class I - III adults of either sex
* Women of childbearing potential must be currently practicing an acceptable form of birth control, and have a negative urine pregnancy test

Exclusion Criteria

* Patients with known allergy, hypersensitivity or contraindications to anesthetic or analgesic medications
* Patients with clinically-significant medical conditions, such as brain, heart, kidney, endocrine, or liver diseases, peptic ulcer disease or bleeding disorders
* Pregnant or lactating women
* Subjects with a history of alcohol or drug abuse within the past 3 months
* Any other conditions or use of any medication which may interfere with the conduct of the study (e.g., asthmatic patients history of asthma, chronic cough, or upper respiratory tract infection during the previous 2 wk or recent treatment with angiotensin-converting enzyme inhibitors, bronchodilators, or steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Wender, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States

REFERENCES:
- [Derived] White PF, Elvir-Lazo OL, Zaentz AS, Kariger R, Yumul R, Khany MM, Stern A, Vuong M, Wender RH. Does small-dose fentanyl improve perioperative outcomes in the ambulatory setting? A randomized, double-blind, placebo-controlled study. Acta Anaesthesiol Scand. 2015 Jan;59(1):56-64. doi: 10.1111/aas.12424. Epub 2014 Oct 20. PMID 25329822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to the day of surgery, potential study patients scheduled to undergo superficial surgical procedures received a packet of materials from their surgeon. The packet contained an initial patient contact letter, a privacy information sheet, and the institution review board (IRB)-approved informed consent form.
Period: Overall Study
Arm/Group | Fentanyl | Saline Solution
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl: Fentanyl (50 µg/ml) 2 ml at induction, 1-2 ml boluses as needed
  Saline: 2 ml at induction 1-2 ml boluses as needed
- Saline Solution: Saline Solution 2 ml at induction, 1-2 ml boluses as needed
  Fentanyl: Fentanyl (50 µg/ml) 2 ml at induction, 1-2 ml boluses as needed
- Total: Total of all reporting groups
Arm/Group | Fentanyl | Saline Solution | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (14) | 48 (16) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Coughing
Description: during the perioperative period (insertion of an LMA device, maintenance of anesthesia, and emergence from general anesthesia) for ambulatory surgery procedures.
Time Frame: one day
Measure: Number; unit: participants
Arm/Group | Fentanyl | Saline Solution
Number analyzed (Participants) | 50 | 50
participants | 10 | 6

2. Secondary Outcome: Incidence of Nausea and Vomiting
Description: Postoperative nausea and vomiting using a Verbal Rating Scale (0-10) at PACU (post-anesthesia care unit.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Fentanyl | Saline Solution
Number analyzed (Participants) | 50 | 50
participants | 2 | 4

3. Secondary Outcome: Postoperative Pain
Description: Postoperative pain measured using a Verbal Rating Scale (VRS) at post-anesthesia care unit (PACU), (90 minutes after arriving).
  Postoperative pain VRS scores: 0 = none pain to 10 = intolerable pain.
Time Frame: one day
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fentanyl | Saline Solution
Number analyzed (Participants) | 50 | 50
Scores on a scale | 1.5 (1.8) | 1.5 (1.6)

ADVERSE EVENTS:
Time Frame: No adverse event reported during the study period.
Arm/Group | Fentanyl | Saline Solution
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No